CLINICAL TRIAL: NCT02086942
Title: Randomized, Multicenter Study of Tolerability and Efficacy of Modified Combinations of Bortezomib, Dexamethasone and Cyclophosphamide in Previously Untreated Multiple Myeloma.
Brief Title: Tolerability and Efficacy of Modified VCD Regimens in Previously Untreated Multiple Myeloma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yongping Zhai (Other)
Responsible Party: Sponsor-Investigator, Yongping Zhai, Department of hemotology, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAB20130806
Record Dates: First submitted 2014-03-12; First posted 2014-03-13 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- modified VCD regimen1 (Experimental): Induction therapy：modified VCD regimen1 for 4 cycles,28 Days per Cycle.Intensive therapy：modified VCD regimen1 for 5 cycles.
  Maintenance treatment:CP for 12 cycles. Interval between every two cycles for one month.
  Interventions:
  Drug: Bortezomib 1.6mg/m2 SC,Days 1, 6, 11, 16; Drug:Cyclophosphamide 300mg/m2 VD,Days 1-3; Drug: Dexamethasone 40 mg/d VD,Days 1, 6, 11,16; We undertook a pharmacodynamic substudy at selected sites. Blood samples were collected in cycle 1 on day 1, 6,11,16 before the dose was given and at several time points after dosing. We analysed whole blood samples to measure 20S proteasome chymotryptic activity, with a standard method. Pharmacodynamic parameters were calculated by analysis of percentage inhibition of 20S proteasome activity-time data.
  Interventions: Drug: Bortezomib; Drug: cyclophosphamide; Drug: Dexamethasone
- modified VCD regimen2 (Experimental): Induction therapy：modified VCD regimen1 for 4 cycles,28 Days per Cycle.Intensive therapy：modified VCD regimen 2 for 5 cycles.
  Maintenance treatment:CP for 12 cycles. Interval between every two cycles for one month.
  Interventions:
  Drug: Bortezomib 1.3mg/m2 SC,Days 1, 6, 11, 16; Drug:Cyclophosphamide 300mg/m2 VD,Days 1-3; Drug: Dexamethasone 40 mg/d VD,Days 1, 6, 11,16; We undertook a pharmacodynamic substudy at selected sites. Blood samples were collected in cycle 1 on day 1, 6,11,16 before the dose was given and at several time points after dosing. We analysed whole blood samples to measure 20S proteasome chymotryptic activity, with a standard method. Pharmacodynamic parameters were calculated by analysis of percentage inhibition of 20S proteasome activity-time data.
  Interventions: Drug: Bortezomib; Drug: cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Induction therapy：1.6mg/m2 or 1.3mg/m2 SC,Days 1, 6, 11, 16 of each 28 day cycles,4 cycle Intensive therapy：1.6mg/m2 or 1.3mg/m2 SC,Days 1, 6, 11, 16 of each 28 day cycles,5 cycles.
  Other Names: Velcade
Drug: cyclophosphamide — Induction therapy：300mg/m2 VD Days 1-3 of each 28 day cycles,4 cycles. Intensive therapy：300mg/m2 VD Days 1-3 of each 28 day cycles,5 cycles. Maintenance treatment with CP: 200mg PO Days 1-14 of each 28 day cycles,12 cycles.
  Other Names: Endoxan, Cytoxan, Neosar, Procytox, Revimmune
Drug: Dexamethasone — Induction therapy：40 mg/d VD Days 1,6,11,16 of each 28 day cycles,4 cycles Intensive therapy：40 mg/d VD Days 1,6,11,16 of each 28 day cycles,5 cycles.
  Other Names: Acidocont,Deronil,Dexacortal,dexametona,Flumeprednisolon

SUMMARY:
This phase 2 study will be conducted at 10 centers and enroll patients from August 2013 to August 2017.Firstly, All patients included will provide written informed consent. Secondly, they will be randomized equally to receive modified VCD regimen arm 1 or modified VCD regimen arm 2. In total, 47 patients per arm (or 94 in total) are required. The treatment consists of four 4-week cycles of induction therapy followed by intensive therapy with another five modified VCD regimens and maintenance treatment with CP regimen. Then, patients will be followed up for 24 months after chemotherapy. The investigators will record all the laboratory and clinical investigations to assess response at different points of the study. We also monitor and assess adverse events (AEs), as graded according to NCI-CTCAE Version 3.0.Response categories were based on the International Myeloma Working Group uniform response criteria.In addition, 20 patients (10 in VCD regimen arm 1 group, 10 in VCD regimen arm 2 group) from ten centres will be enrolled in the pharmacodynamic substudy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated symptomatic MM
* 18 years of age or older, regardless of gender
* secretory MM with measurable diseases
* Karnofsky Performance Status≥50%（pathological fractures excluded）
* Patients without heart and pulmonary dysfunction ≤class I

Exclusion Criteria:

* peripheral neuropathy of grade 2 or higher according to NCI-CTCAE Version 3.0
* Relapse and refractory MM
* MM without symptom
* Non-secretory MM without measurable diseases
* Karnofsky Performance Status<50%（pathological fractures excluded）
* Patients with heart and pulmonary dysfunction> class I

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
the rate of complete remission | Day 1 of every treatment cycle
  The rate of complete remission of modified VCD regimens in patients with MM assessed by International Myeloma Working Group(IMWG) criteria.

SECONDARY OUTCOMES:
progression free survival | up to two year
  PFS of modified VCD regimens in patients with MM assessed by International Myeloma Working Group(IMWG) criteria.
Adverse Events | up to two years
  Adverse events (AEs) were graded according to NCI-CTCAE Version 4.0
overall response rates (ORR) | Day 1 of every treatment cycle
  The rate of overall response of modified VCD regimens in patients with MM assessed by International Myeloma Working Group(IMWG) criteria.
duration of response | up to 6 months
  Duration of response of modified VCD regimens in patients with MM assessed by International Myeloma Working Group(IMWG) criteria.
overall survival (OS) | up to two year
  The rate of OS of modified VCD regimens in patients with MM assessed by International Myeloma Working Group(IMWG) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: zhai yo ping, doctor, Principal Investigator — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li F, Yao FS, Zhu XJ, Gu WY, Wang XH, Chen B, Huang DP, Ding JH, Wu TQ, Zhu Y, Zhao Q, Tang YM, Song P, Zhou XG, An ZM, Guo X, Wang XL, Zhong L, Xie XB, Zhai YP. A randomized phase II, open-label and multicenter study of combination regimens of bortezomib at two doses by subcutaneous injection for newly diagnosed multiple myeloma patients. J Cancer Res Clin Oncol. 2019 Sep;145(9):2343-2355. doi: 10.1007/s00432-019-02967-3. Epub 2019 Jul 6. PMID 31280348